CLINICAL TRIAL: NCT06786364
Title: Types of Photoplethysmographic Waves in Adult Patients with Septic Shock
Acronym: SHOCK PLETH
Status: Recruiting | Type: Observational
Sponsor: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Juan Fernando Bautista Garcia, MD, Hospital General de México Dr. Eduardo Liceaga
Other Study IDs: DI/24/401/03/33
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Shock Septic; Photoplethysmography; Waveform
Keywords: shock septic; waveform; vasodilation; Photoplethysmography; arterial tone
MeSH Terms: conditions — Shock, Septic; Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this study is to identify the types of Photoplethysmographic waves present in adults with septic shock and determine whether these waves correlate with other variables of tissue hypoperfusion such as capillary refil, serum lactate and mottling score.

DETAILED DESCRIPTION:
Photoplethysmography is the technology used in pulse oximeters in order to calculate arterial oxygen saturation and pulse rate, this technology generates a wave whose morphology has been related to blood flow and arterial tone. Recently Tusman and collaborators described a morphological classification of the photoplethysmografic wave that has a high correlation with arterial tone, such classification is divided in 6 types; Types I and II indicate vasoconstriction, Type III normal arterial tone and Types IV, V and VI describe mild, medium and severe vasodilation respectively, therefore it could be used to identify the arterial tone in those patients with septic shock. This study will identify the type of photoplethysmographic waves that are present in adults with septic shock based in the Tusman and collaborators classification, it will also describe the frequency of appearance and their correlation with other hemodynamic variables such as capillary refill, serum lactate, mottling score, heart rate, mean arterial pressure, pulse pressure and perfusion index.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of 18 years of age and above dignossed with septic shock according to the definition stated in Sepsis 3.0
* Patients with axillary temperature above 36°C
* Patients and/or family that agree to participate in such study and sign the informed consentment
* Patients that tolerate supine position

Exclusion Criteria:

* Patients with Cardiogenic shock, hipovolemic, obstructive and distributive (neurogenic, anafilactic) shock the exception being septic shock
* Patients with history of any type of cardiac arrhythmia
* Patients with history of chronic hepatic disease
* Patients with limited or diffuse systemic sclerosis
* Patients that have scarring, nail polish or thickened nails that may impede the proper placement and accurate measurement of photoplethysmography with the pulse oximeter
* Patients with history of heart insufficiency P- atients with septic shock that already have vasopressor aggents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the emergency department at "Hospital General de México Dr. Eduardo Liceaga" and meet the criteria for septic shock established in Sepsis 3.0 and have signed the informed consentment will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Photoplethysmography wave types in adult patiens with septic shock | After the inclusion of the patient.
  The type of Photoplethysmography wave obtained and digitized through the sensor of a conventional pulse oximeter without autoscale. The wave will be classified in type I, II, III, IV, V and VI according to the criteria proposed by Tusman and collaborators

SECONDARY OUTCOMES:
Capillary refill | After the inclusion of the patient
  Mesurement of the time it takes for the ventral surface of the fingers to return to its normal color after being compressed by a transparent microscope slide for 10 seconds. Measured in seconds.
Mottling score | After the inclusion of the patient
  Classification regarding the type of mottling surrounding the knee in each patient. The classification is as folllows 0= no mottling, 1= Mottling the size of a coin on the knee, 2= mottling extending just over the superior part of the knee, 3= Mottling covering up to half the thigh, 4= mottling continues to the inguinal fold, 5= severe mottling extending beyond the inguinal area.
Serum lactate levels | After the inclusion of the patient
  Mesurement of serum lactate through venous blood gass analysis at hospital admittanace. Mesured in mmol/L
Heart rate | After the inclusion of the patient
  Determination of the number of heart beats per minute in patients obtenined with telemetry. Messured in beats per minute
Sistolic and diastolic blood pressure | After the inclusion of the patient
  Messurement of arterial blood pressure with an adult sized aneroid sphygmomanometer. Messurement in mmHg.
Perfussion index | After the inclusion of the patien
  Messurement of the perfusion index obtained and calculated by a sensor in a conventional pulse oximeter without autoscale. Measurement in whole numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Fernando Bautista Garcia, MD, Principal Investigator — Hospital General de México Dr. Eduardo Liceaga
Locations (1):
- Hospital General de México Dr. Eduardo Liceaga, Mexico City, Cuauhtemoc, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tusman G, Acosta CM, Pulletz S, Bohm SH, Scandurra A, Arca JM, Madorno M, Sipmann FS. Photoplethysmographic characterization of vascular tone mediated changes in arterial pressure: an observational study. J Clin Monit Comput. 2019 Oct;33(5):815-824. doi: 10.1007/s10877-018-0235-z. Epub 2018 Dec 15. PMID 30554338